CLINICAL TRIAL: NCT02717481
Title: Using Ultrasound to Evaluate Aortic Aneurysm Size Based on 3D Co-registration to Previous Computerized Tomography
Brief Title: Using US to Evaluate Aortic Aneurysm Size Based on 3D Co-registration to Previous CT Scan
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0551-15 RMB CTIL
Record Dates: First submitted 2016-03-13; First posted 2016-03-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with known aortic aneurysm: Patients with known abdominal aortic aneurysm diagnosed in clinical follow-up or after an invasive procedure to repair it.
  US-CT Fusion examination
  Interventions: Device: US-CT Fusion examination

INTERVENTIONS:
Device: US-CT Fusion examination — Patients will undergo an US examination using an US device with US-CT Fusion capabilities.

SUMMARY:
Examine a new method based on fusion between ultrasound (US) and previous ultrasound/computerized tomography(US/CT) studies to evaluate the size of abdominal aneurysm and measure the changes over time and following invasive repair procedure.

DETAILED DESCRIPTION:
Selection test for assessing aortic aneurysm is CT angio, it performed after injection of contrast material and allows a complete demonstration of the blood vessels. This test exposes the patient to ionizing radiation and the injection of iodine contrast medium. Repeated tests pose a risk of developing a malignancy in the future due to the use of ionizing radiation and risk of renal impairment and allergic reactions due to the injection of contrast material. Ultrasound is another test that enables the detection and evaluation of aortic aneurysm. Patients with a known diagnosis of aortic aneurysm detected on CT are required to continuous monitoring in light of its growth over time and the risk of rupture.

Using Co-registration over the US device will enable to conduct a US directed aorta examination, which uses the information produced from the CT as a "roadmap" for detection and localization of the aneurysm. That can theoretically improve detection capabilities and characteristics of the aneurysm and outcomes of the invasive treatment.

ELIGIBILITY:
Inclusion Criteria:

•Patients with abdominal aortic aneurysm diagnosis in clinical follow-up or after an invasive procedure to fix it.

Exclusion Criteria:

* Inability to perform Ultrasound
* Pace maker
* Hemodynamic instability
* Inability to cooperate in US examination
* Pregnant Women - does not undergo CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with abdominal aortic aneurysm diagnosis in clinical follow-up or after an invasive procedure to fix it
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Exact and reliable evaluation of the aneurysm size | two years
  The size of the aneurysm will be evaluated by two different doctors or twice with large time frame between the studies. The difference between the measurements with the fusion technology will be compared to the difference without the fusion technology.
  The accuracy of the measurement will be evaluated by comparing to previous CT examination.

SECONDARY OUTCOMES:
The size difference between systolic and diastolic aneurysm. | two years
Aneurysm neck size and changes following an invasive procedure to repair it (EVAR). | two years
Evaluation of the pressure on the aneurysmal wall. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Diana Gaitini, MD, Prof., Principal Investigator — Director of Ultrasound Unit, Rambam Health Care Campus
Locations (1):
- Rambam healt care campus, Department of Medical Imaging, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Kobeiter H, Nahum J, Becquemin JP. Zero-contrast thoracic endovascular aortic repair using image fusion. Circulation. 2011 Sep 13;124(11):e280-2. doi: 10.1161/CIRCULATIONAHA.110.014118. No abstract available. PMID 21911788
- [Background] McNally MM, Scali ST, Feezor RJ, Neal D, Huber TS, Beck AW. Three-dimensional fusion computed tomography decreases radiation exposure, procedure time, and contrast use during fenestrated endovascular aortic repair. J Vasc Surg. 2015 Feb;61(2):309-16. doi: 10.1016/j.jvs.2014.07.097. Epub 2014 Aug 28. PMID 25175634
- [Background] Pfister K, Schierling W, Jung EM, Apfelbeck H, Hennersperger C, Kasprzak PM. Standardized 2D ultrasound versus 3D/4D ultrasound and image fusion for measurement of aortic aneurysm diameter in follow-up after EVAR. Clin Hemorheol Microcirc. 2016;62(3):249-60. doi: 10.3233/CH-152012. PMID 26484714